CLINICAL TRIAL: NCT06758089
Title: A Clinical Comparison of Two Soft Toric Contact Lenses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-163
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-10

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens 1 (ocufilcon D) (Experimental): All participants will wear lens 1 for 15 minutes (Period 1).
  Interventions: Device: Lens 1 (ocufilcon D)
- Lens 2 (somofilcon A) (Experimental): All participants will wear lens 2 for 15 minutes (Period 2).
  Interventions: Device: Lens 2 (somofilcon A)

INTERVENTIONS:
Device: Lens 1 (ocufilcon D) — 15 minutes of daily wear
  Arms: Lens 1 (ocufilcon D)
Device: Lens 2 (somofilcon A) — 15 minutes of daily wear
  Arms: Lens 2 (somofilcon A)

SUMMARY:
The aim of this study is to compare the short-term clinical performance of two toric contact lenses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the short-term clinical performance of two toric contact lenses when compared to each other after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age and capacity to volunteer.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They currently wear soft contact lenses, or have done so within the past two years.
5. They have ocular astigmatism in both eyes of between 0.75DC and 2.00DC.
6. They have a spherical component: plano to -7.00DS (based on ocular refraction).
7. They are expected to be able to be fitted with the study lenses within the power range available.

Exclusion Criteria:

1. They have an ocular disorder, which would normally contra-indicate contact lens wear.
2. They have a systemic disorder, which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or breastfeeding.
8. They have an eye or health condition including an immunosuppressive or infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or a history of anaphylaxis or severe allergic reaction.
9. They have taken part in any contact lens or care system clinical research within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Overall Score | At the end of 15 minutes of daily wear
  The primary outcome measure for this study is the subjective overall score on a scale of 0-100 (0= Extremely poor, unmanageable, cannot use lenses, 100= Excellent, highly impressed with these lenses overall).

SECONDARY OUTCOMES:
Subjective Vision | At the end of 15 minutes of daily wear
  The secondary outcome measure for this study is the subjective vision on a scale of 0-100 (0= Extremely poor, intolerable, lenses cannot be worn, 100= Excellent, unaware of any visual loss).
Subjective Comfort | At the end of 15 minutes of daily wear
  The secondary outcome measure for this study is the subjective comfort on a scale of 0-100 (0= Extremely uncomfortable, causes pain, cannot be tolerated, 100= Excellent, cannot be felt).

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codina, PhD, FBCLA, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom